CLINICAL TRIAL: NCT02348619
Title: A Six-Week, Double-Blind, Placebo-Controlled, Randomized- Withdrawal, Multicenter Study of the Safety and Efficacy of JZP-110 [(R)-2-amino-3-phenylpropylcarbamate Hydrochloride] in the Treatment of Excessive Sleepiness in Subjects With Obstructive Sleep Apnea (OSA)
Brief Title: "Six-week Study of the Safety and Efficacy of JZP-110 in the Treatment of Excessive Sleepiness in OSA"
Acronym: OSA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-004
Record Dates: First submitted 2015-01-15; First posted 2015-01-28 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — solriamfetol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 75, 150, 300 mg of JZP-110 (Active Comparator): Once Daily Dosing
  Interventions: Drug: JZP-110
- Placebo (Active Comparator): Once Daily Dosing
  Interventions: Drug: JZP-110

INTERVENTIONS:
Drug: JZP-110

SUMMARY:
This trial is a 6-week, double-blind, placebo-controlled, randomized-withdrawal, multicenter study of safety and efficacy of JZP-110 in the treatment of excessive sleepiness in adult subjects with OSA.

ELIGIBILITY:
Major Inclusion Criteria:

1. Male or female between 18 and 75 years of age, inclusive
2. Diagnosis of OSA according to ICSD-3 criteria
3. Body mass index from 18 to <45 kg/m2
4. Consent to use a medically acceptable method of contraception
5. Willing and able to provide written informed consent

Major Exclusion Criteria:

1. Female subjects who are pregnant, nursing, or lactating.
2. Any other clinically relevant medical, behavioral, or psychiatric disorder other than OSA that is associated with excessive sleepiness
3. History or presence of bipolar disorder, bipolar related disorders, schizophrenia, schizophrenia spectrum disorders, or other psychotic disorders according to DSM-5 criteria
4. History or presence of any acutely unstable medical condition, behavioral or psychiatric disorder (including active suicidal ideation), or surgical history that could affect the safety of the subject or interfere with study efficacy or safety assessments or the ability of the subject to complete the trial per the judgment of the principal investigator
5. History of bariatric surgery within the past year or a history of any gastric bypass procedure
6. Presence or history of significant cardiovascular disease
7. Use of any over the counter (OTC) or prescription medications that could affect the evaluation of excessive sleepiness
8. Received an investigational drug in the past 30 days or five half-lives (whichever is longer)
9. Previous exposure to or participation in a clinical trial of JZP-110 (ADX-N05, R228060, or YKP10A)
10. History of phenylketonuria (PKU) or history of hypersensitivity to phenylalanine-derived products

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (22):
  - Sleep Disorder Center of Alabama, Birmingham, Alabama
  - The Research Center of Southern California, Oceanside, California
  - SDS Clinical Trials, INC, Orange, California
  - Santa Monica Clinical Trials, Santa Monica, California
  - Critical Care Pulmonary & Sleep Associates, LLC, Lakewood, Colorado
  - PAB Clinical Research, Brandon, Florida
  - Broward Research Group, Inc., Hollywood, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - Emory Sleep Center, Atlanta, Georgia
  - Rowe Neurology Institute RNI - Lenexa, Lenexa, Kansas
  - Veritas Clinical Specialities LTD, Topeka, Kansas
  - Advanced Neurodiagnostic Ceneter, Metairie, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham & Womens Hospital, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Center for Sleep & Circadian Neurobiology, Philadelphia, Pennsylvania
  - UPMC Sleep Medicine Center, Pittsburgh, Pennsylvania
  - Lowcountry Lung Critical Care, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - EVMS Sleep Medicine, Norfolk, Virginia
  - American Sleep Medicine, Vienna, Virginia
- Finland (3):
  - Tampere University Hospital, Tampere, Södra Finlands Län
  - Turku University Hospital, Sleep Clinic, Turku, Västra Finlands Län
  - Helsinki Sleep Center, Helsinki
- France (2):
  - Grenoble University Hospital, La Tronche, Auvergne-Rhône-Alpes
  - CHU de Poitiers, Poitiers, Vienne
- Germany (2):
  - Klinische Forschung Schwerin GmbH, Schwerin, Mecklenburg-Vorpommern
  - Somnolab Dortmund, Dortmund, North Rhine-Westphalia
- Department of Sleep Medicine, Gӧteborg, Västra Götaland County, Sweden

REFERENCES:
- [Derived] Strollo PJ Jr, Hedner J, Collop N, Lorch DG Jr, Chen D, Carter LP, Lu Y, Lee L, Black J, Pepin JL, Redline S; Tones 4 Study Investigators. Solriamfetol for the Treatment of Excessive Sleepiness in OSA: A Placebo-Controlled Randomized Withdrawal Study. Chest. 2019 Feb;155(2):364-374. doi: 10.1016/j.chest.2018.11.005. Epub 2018 Nov 22. PMID 30471270

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following screening, subjects entered the Titration phase. Subjects who were titrated to an efficacious and tolerable dose in the Titration phase remained on the same dose regimen in the Stable-Dose phase. Subjects in the Double-Blind Withdrawal phase who did not receive JZP-110 received placebo for 2 weeks.
Groups:
- JZP-110: Start at 75 mg, titrate up to 150 or 300 mg, or down at any time.
- Placebo: Subjects in the Double-Blind Withdrawal phase who did not receive JZP-110 received placebo for 2 weeks.
Period: Titration Phase
Arm/Group | JZP-110 | Placebo
Started | 174 | 0
Completed | 157 | 0
Not Completed | 17 | 0
Period: Stable-Dose Phase
Arm/Group | JZP-110 | Placebo
Started | 157 | 0
Completed | 124 | 0
Not Completed | 33 | 0
Period: Double-Blind Withdrawal Phase
Arm/Group | JZP-110 | Placebo
Started | 62 | 62
Completed | 60 | 62
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Double-Blind Withdrawal Phase
Number analyzed (Participants) | 124
Age, Continuous [Mean (Standard Deviation); unit: years]
  Placebo | 56.2 (9.75)
  JZP-110 | 56.3 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: A total of 124 subjects were randomized into the Double-Blind Withdrawal phase of the study and comprised the Safety population for that phase. Two of these subjects were excluded.
  Participants
    Placebo: number analyzed (Participants) | 62
    Placebo: Female | 21
    Placebo: Male | 41
    JZP-110: number analyzed (Participants) | 62
    JZP-110: Female | 26
    JZP-110: Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total of 124 subjects were randomized into the Double-Blind Withdrawal phase of the study and comprised the Safety population for that phase. Two of these subjects were excluded.
  Participants
    Placebo: number analyzed (Participants) | 62
    Placebo: American Indian or Alaska Native | 0
    Placebo: Asian | 2
    Placebo: Native Hawaiian or Other Pacific Islander | 0
    Placebo: Black or African American | 15
    Placebo: White | 45
    Placebo: More than one race | 0
    Placebo: Unknown or Not Reported | 0
    JZP-110: number analyzed (Participants) | 62
    JZP-110: American Indian or Alaska Native | 0
    JZP-110: Asian | 0
    JZP-110: Native Hawaiian or Other Pacific Islander | 0
    JZP-110: Black or African American | 12
    JZP-110: White | 50
    JZP-110: More than one race | 0
    JZP-110: Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in the Maintenance of Wakefulness Test (MWT)
Description: Change in the mean sleep latency time as determined from the first four trials of a 40-minute MWT from the end of the Stable Dose Phase to the end of the Double-blind Withdrawal Phase. Mean sleep latency defined as the average of the first four MWT trial's measurements.
Time Frame: Week 4 to Week 6
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | JZP-110 | Placebo
Number analyzed (Participants) | 60 | 62
minutes | -0.96 (1.350) | -12.11 (1.326)

2. Primary Outcome: Change in the Epworth Sleepiness Scale (ESS)
Description: Change in Epworth Sleepiness Scale (ESS) score from the end of the Stable Dose Phase to the end of the Double-blind Withdrawal Phase. A negative change from baseline represents improvement in excessive sleepiness.
  The ESS is a self-administered questionnaire with 8 questions. Each activity is scored on a scale ranging from 0-3, with 0 = would never fall asleep, and 3 = high chance of falling asleep. The total score ranges from 0-24, with a higher number representing an increased propensity for sleepiness. An analysis of covariance (ANCOVA) was used for the analysis of ESS scores. The response variable was the change in ESS score from week 4 to week 6.
Time Frame: Week 4 to Week 6
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | JZP-110 | Placebo
Number analyzed (Participants) | 60 | 62
points on a scale | -0.1 (0.73) | 4.5 (0.71)

3. Secondary Outcome: Patient Global Impression of Change (PGIc)
Description: Percentage of subjects reported as worse (minimally, much, or very much) on the PGIc at the end of the Double-blind Withdrawal Phase. PGIc was rated by subjects and measures the change in their condition since treatment starts on a 7-point scale ranging from 1= very much improved to 7= very much worse.
Time Frame: Week 4 to Week 6
Measure: Number; unit: percentage of subjects
Arm/Group | JZP-110 | Placebo
Number analyzed (Participants) | 60 | 62
percentage of subjects | 20 | 50

4. Secondary Outcome: Clinical Global Impression of Change (CGIc)
Description: Percentage of subjects reported as worse (minimally, much, or very much) on the CGIc at the end of the Double-blind Withdrawal Phase. CGIc was rated by clinicians and measures the change in the subject's condition since treatment starts on a 7-point scale ranging from 1= very much improved to 7= very much worse.
Time Frame: Week 4 to Week 6
Measure: Number; unit: percentage of subjects
Arm/Group | JZP-110 | Placebo
Number analyzed (Participants) | 60 | 62
percentage of subjects | 22 | 59

5. Secondary Outcome: Change in Functional Outcomes of Sleep Questionnaire (FOSQ-10)
Description: Change is total score from the end of the stable dose phase to the end of the double blind withdrawal phase. Functional Outcomes of Sleep Questionnaire Short Version (FOSQ-10) is a 10-item disease-specific quality of life questionnaire to assess the effect of excessiveness sleepiness on multiple activities of everyday living. The FOSQ-10 consists of 10 questions, each scored on a scale from 1-4. The questionnaire has a 4-point response format for each question (1 = extreme difficulty, 2 = moderate difficulty, 3 = a little difficulty, and 4 = no difficulty). The total score is derived by the mean of the 5 subscale scores, multiplied by 5, resulting in a possible range of scores between 5 to 20; lower FOSQ-10 scores are worse, indicating more difficulty carrying out activities; higher FOSQ-10 scores are better, indicating less difficulty carrying out activities.
Time Frame: Week 4 to Week 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | JZP-110 | Placebo
Number analyzed (Participants) | 60 | 62
units on a scale | -0.15 (0.393) | -1.31 (0.381)

ADVERSE EVENTS:
Groups:
- JZP-110 (Entire Study): Across the entire study.
- Placebo (Randomized Withdrawal): During the randomized withdrawal phase only.
Arm/Group | JZP-110 (Entire Study) | Placebo (Randomized Withdrawal)
All-Cause Mortality (participants affected / at risk) | 0/174 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/174 | 0/62
Other Adverse Events (participants affected / at risk) | 58/174 | 0/62
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | JZP-110 (Entire Study) (N=174) | Placebo (Randomized Withdrawal) (N=62)
Headache (Nervous system disorders) | 20 | 0
Dizziness (Nervous system disorders) | 14 | 0
Dry mouth (Gastrointestinal disorders) | 13 | 0
Nausea (Gastrointestinal disorders) | 13 | 0
Insomnia (Psychiatric disorders) | 11 | 0
Palpitations (Cardiac disorders) | 9 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review trial results communications prior to public release and can embargo such communications for a period of at least 60 days from the time submitted to sponsor for review. If requested by sponsor, the PI will withhold publication for up to an additional 30 days. Furthermore, the first publication of study results must be a joint publication of all study sites unless a joint manuscript has not been submitted for publication within 12 months of completion of the study.

DOCUMENTS (2):
  • Study Protocol (2016-02-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT02348619/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT02348619/SAP_001.pdf